STUDY PROTOCOL FOR EVALUATE THE EFFECTIVENESS OF PROGESTIN-PRIMED VERSUS GNRH ANTAGONIST PROTOCOLS IN VIETNAMESE WOMEN UNDERGOING IN-VITRO FERTILIZATION

**PROTOCOL ID: 9720105** 

**DOCUMENT DATE: December 15, 2023** 

Author list: Than Trong Thach<sup>1\*</sup>, Le Duc Thang<sup>2</sup>, Nguyen Ha Ngoc Thien Thanh<sup>3</sup>, Duong Thi Ngoc Chau<sup>1</sup>, Le Thai Thanh Khue<sup>1</sup>, Nguyen Manh Ha<sup>4</sup>, Le Hoang<sup>2</sup>

Affiliation: <sup>1</sup>University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam; <sup>2</sup>Tam Anh General Hospital, Hanoi, Vietnam; <sup>3</sup>An Sinh Hospital, Ho Chi Minh City, Vietnam; <sup>4</sup>IVF and Tissue Engineering Center, Hanoi Medical University Hospital, Hanoi, Vietnam

Corresponding author: Thach Than Trong

Email: thachthan007@gmail.com

ORCID ID: <u>0000-0003-1746-7267</u>

Phone: +84908400040

Address: Binh Thanh District, Ho Chi Minh City, Vietnam

#### **BACKGROUND**

Controlled Ovarian Stimulation (COS) plays a significant role in the cycle of In Vitro Fertilization (IVF) or Intra-Cytoplasmic Sperm Injection (ICSI). Premature luteinizing hormone (LH) surge is the main reason for cycle cancelation during COS (1). Two principal methods of pituitary suppression are employed to delay the onset of LH peak in the COS cycle: (1) prolonging the administration of a gonadotropin-releasing hormone agonist (GnRH-a) before the implementation of COS in a long-acting agonist regimen (2) immediate pituitary suppression with a gonadotropin-releasing hormone antagonist (GnRH-ant) in a short-acting antagonist regimen (2). Recently, with the successful development of embryo freezing and thawing techniques, a new COS protocol was proposed using progestin as a "primer" (Progestin-Primed Ovarian Stimulation – PPOS) in the act of inhibiting the LH peak and preventing ovulation occurrence. In 2015, Kuang et al. first reported this protocol and demonstrated efficacy in preventing premature luteinization (3). The PPOS protocol is dominant due to its patient-friendly benefits: oral administration, convenience, and lower cost. Several studies have highlighted the potency of PPOS in prohibiting premature LH surge and promoting positive pregnancy outcomes compared to classical COS regimens in infertile women with normal ovarian reserve (NOR) or those with polycystic ovary syndrome (PCOS) (4-11).

An important factor in determining the effect of progesterone (stimulatory or inhibitory) on pre-ovulatory gonadotrophin secretion, or even its synergistic or antagonistic effect with estrogen, is the timing of administration, the rate of administration, and P4/E2 hormone ratio. Previous studies still have not had consensus; some studies show that at the end of the follicular phase, progesterone concentration increases slightly due to the secretion of granulosa cells of pre-ovulatory antral follicles, causing a slight increase in LH concentration, proving the role of progesterone's stimulating role on gonadotropins (12); However, the LH peak only achieve when progesterone is administered after estrogen has previously been primed. On the other hand, high levels of progesterone from early in the menstrual cycle have been shown to suppress LH peaking (13), with its primary role being

to inhibit follicle development and subsequent inhibition of ovulation, which is the contraceptive basis of progestin-only contraceptives. Recently, it has not been possible to use a single hypothesis related only to estradiol, progesterone, gonadotrophin, GnRH, kisspeptin, and the time to start taking progestogen to explain the mechanism of LH peak appearance and ovulation induction. DYG is a potential alternative progestin for the PPOS protocol in ART (4, 10); it has a high selectivity for progesterone receptors with potent progestogenic activity. In contrast to other progestins, DYG has no clinically relevant agonistic or antagonistic action on the androgen, estrogen, and glucocorticoid receptors and only mild antimineralocorticoid features. Unlike natural progesterone, dydrogesterone has good oral bioavailability; therefore, it may reduce the side effects of progestins (14-16). However, few studies compared the PPOS protocol's efficacy with DYG and GnRH-antagonist protocols. In this RCT, we compared the effects of two protocols, PPOS using DYG and GnRH-ant, on the ovarian response and clinical outcomes in patients undergoing IVF or ICSI.

#### **METHODS AND ANALYSIS**

#### Objectives

This trial aims to compare the efficacy and safety of the PPOS protocol to the GnRH antagonist protocol in patients undergoing IVF procedures.

#### Design of the trial

This was an open-label, randomized controlled trial conducted at the Assisted Reproduction Center of Tam Anh General Hospital between January 2023 and December 2024. The study aimed to estimate the efficacy of the intervention (PPOS protocol) compared to a control group receiving a gonadotropin-releasing hormone (GnRH) antagonist protocol. Inclusion criteria were women aged 20-45 years undergoing IVF. Exclusion criteria included failure to complete ovarian stimulation, systemic diseases like renal failure or lupus, uterine abnormalities, random-start controlled ovarian stimulation cycles, and preimplantation genetic testing for aneuploidies. The study details were explained to all participants, and informed consent was provided. This study was approved

by the Ethics Committee of Hanoi Medicine University, decision number 842, dated July 7, 2023.

#### Eligibility criteria

Eligible patients must meet all inclusion criteria, and no listed exclusion criteria exist.

#### **Inclusion criteria**

Women meeting the sample selection criteria are as follows: (1) Women aged 20 to 45; (2) Infertility due to male factors, fallopian tube factors, or unknown causes; (3) Undergoing IVF in one COS cycle and intended to apply either GnRH antagonist protocol or PPOS protocol; (4) Voluntary participation in research.

#### **Exclusion criteria**

Women who met any of the following criteria were excluded: (1) Any contraindications to ovarian stimulation and IVF/ICSI treatment; (2) Hyperprolactinemia or other endocrine diseases; (3) Those who took hormone drugs within the past three months; (4) Suffering from systemic diseases such as kidney failure, lupus erythematosus, depression, etc.; (5) Abnormal structure of the uterine cavity; (6) Patients with endometriosis or cancer; (7) Random-start cycles; (8) Oocyte donation cycles; (9) Perform embryo biopsy.

#### Recruitment of study participants

Infertile patients come for examination at the Assisted Reproduction Center of Tam Anh General Hospital, Hanoi, and the Assisted Reproduction and Graft Technology Center of Hanoi Medical University. In the basic infertility examination process at the hospital, the clinicians will consider the patient's inclusive and exclusive criteria. The clinicians will contact a research team member if the inclusive criteria are met. A research team member or hospital physician will invite the patient to participate, advise on the study procedure and the benefits and risks of participating, and answer any patient questions (Appendix 2). If the patients agree to participate, they will consent to participate in the trial (Appendix 3). Each participant will be randomly assigned to the treatment group using the PPOS protocol or the control group using the GnRH-ant regimen.

#### Sample size estimation

The sample size was estimated to optimize the precision of non-inferiority testing. This statistical inference is based on a Negative Binomial (NBI) regression model, which aims to compare the average number of retrieved oocytes (or MII oocytes) between two distinct groups, as described by Cundill and Alexander (2015) (17). The following formula encapsulates the estimation process:

$$\sqrt{N} = \frac{Z_{1-\alpha\sqrt{\left(\frac{1}{\mu_0} + \frac{1}{k_0}\right)\left(\frac{1}{Q_1} + \frac{1}{Q_0}\right)} + Z_{1-\beta\sqrt{\frac{1}{Q_1}\left(\frac{1}{\mu_1} + \frac{1}{k_-1}\right)} + \frac{1}{Q_0}\left(\frac{1}{\mu_0} + \frac{1}{k_0}\right)}}{\log(\mu_0) - \log(\mu_1) - \delta}$$

Where:

N represents the aggregate sample size, with each unit being a cycle or patient.

 $\mu_0$  and  $\mu_1$  denote the average outcome values in the control group (GnRH\_ant regimen) and treatment group (PPOS regimen), respectively. The outcome might be the count of retrieved oocytes or MII oocytes.

 $Q_0$  and  $Q_1$  are the allocation ratios for the control and treatment groups, respectively. They represent the proportion of the total sample size that should be allocated to each group. In our research, both Q0 and Q1 were set to 0.5.

 $k_0$  and  $k_1$  are the dispersion parameters of the NBI distribution for the control and treatment groups, respectively.

 $\delta$  is the non-inferiority margin (in log scale), signifying the minimum clinically or practically significant difference.

 $\mathbb{Z}_p$  is the critical value, or pth percentiles of a standard normal distribution

 $\alpha$  is the Type I error, set at 0.05, and  $\beta$  is the Type II error, set at 0.2 (corresponding to a statistical power of 0.8).

From January 1st to October 10th, 2022, at Tam Anh Hospital, 804 patients underwent ovarian stimulation. We observed average retrieved oocyte counts of 11.2 and 11.4 and average mature oocyte counts of 7.62 and 7.54 in the PPOS and GnRH-ant groups, respectively. We engaged in a simulation process with these observations, utilizing the formula to determine potential sample size values. We let  $\mu 0$  and  $\mu 1$  span an interval from 6 to 12 units, while the difference between the groups ranged from -1.5 to 1.5 units. The non-inferiority margin remained constant at log(1.5) units. The results from this simulation are illustrated in Figure 1. According to this result, we concluded that a sample comprising 200 patients (split equally between the groups) would be required. This size ensures that no difference in the number of retrieved or MII oocytes between the PPOS and control group would exceed 1.5 units.

#### **Randomization Process**

We apply a stratified randomization process to ensure unbiased allocation of participants to GnRH-ant and PPOS treatment arms. The process is designed and executed using Python programming language. Initially, each participant will be assigned a unique identification (ID) constructed from a combination of uppercase letters (A-Z) and numbers (0-9), with customizable ID lengths. Concurrently, each participant is categorized based on the "POSEIDON" criterion, a categorical stratification variable with four potential categories: P1, P2, P3, and P4. Participants are allocated to these strata by a predefined probability distribution of 14.86%, 25.39%, 15.99%, and 43.76%, respectively. This distribution was derived from the actual distribution of POSEIDON categories among patients who underwent IVF treatment at Tam Anh Hospital during 2020-2022. Within each "POSEIDON" stratum, participants are randomized equally across the two treatment groups (GnRH-ant or PPOS protocol). The process ensures that if there's an odd number of units in a stratum, the extra unit is randomized within the stratum rather than across the entire dataset.

#### **Treatment method**

#### Ovarian stimulation protocols

Controlled ovarian hyperstimulation commenced on the second day of the menses utilizing recombinant follicle-stimulating hormone (Follitrope, LG Chem, South Korea) at dosages between 150-300 international units (IU) per day. Initial gonadotropin dosages were determined per patient based on baseline parameters, including age, AMH, baseline FSH, body mass index (BMI), antral follicle count (AFC), and titrated subsequently per folliculogenesis response. In the gonadotropin-releasing hormone (GnRH) antagonist protocol group, pituitary suppression began on stimulation day six via daily 0.25 milligram GnRH antagonist administration (ganirelix or cetrorelix). In the progestin-primed ovarian stimulation (PPOS) group, 30mg/day of dydrogesterone was initiated on cycle day 2 through to trigger day. Serum luteinizing hormone (LH) levels were quantified on stimulation days one, six, and eight alongside trigger day using competitive electrochemiluminescence immunoassays via Cobas analyzer. Once dominant follicles reached  $\geq 20$  mm diameter or  $\geq 3$  follicles met 18 mm threshold, final oocyte maturation was induced. Depending on ovarian hyperstimulation risk, either 0.2 mg triptorelin (Diphereline, Ipsen Pharma Biotech, France) alone was administered for high-risk patients or a Dual trigger consisting of 2000 IU hCG (IVF-C, LG Chem, South Korea) combined with 0.2 mg triptorelin (Diphereline, Ipsen Pharma Biotech, France) was used for the remaining patients. Oocyte retrieval via transvaginal aspiration was performed approximately 36 hours later.

#### Laboratory protocol

Oocyte-cumulus complexes were incubated for 2 hours in G-IVF medium (Vitrolife) using Origio benchtop incubators to complete nuclear maturation. After removing cumulus cells, denuded oocytes were evaluated under an inverted microscope to validate the achievement of metaphase II status, while degenerate, large, or severely dysmorphic oocytes were excluded. Intracytoplasmic sperm injection (ICSI) was executed 3-4 hours post-retrieval by experienced embryologists. Resultant zygotes were cultured in continuous single media

(Fujifilm Irvine Scientific) within tri-gas incubators (37°C, 5% O2, 6% CO2) until day 3. Strict morphological criteria were enforced, only retaining normally fertilized two pronuclei zygotes while eliminating abnormal multinuclear embryos. Cleavage-stage quality was graded at 67-69 hours per Istanbul consensus based on cell number, fragmentation, multinucleation, and uniformity. On post-ICSI day 3, embryologists counseled patients on pursuing blastocyst culture versus cryopreservation. The morphology of the blastocysts was evaluated using the Gardner and Schoolcraft grading system, and embryos meeting the criteria of 3-6 AA/AB/BA blastocysts or 1-2 AA/AB embryos were classified as good quality.

#### **Outcome measurements**

#### Primary outcomes

The primary outcome is the success rates, including maturation, fertilization, and probabilities of achieving Day 3 and Day 5 embryos.

#### Secondary outcomes

The secondary outcome is the process of the evolution of LH levels in the PPOS group.

We transferred the cryopreserved embryo in the next cycle after the stimulation cycle. Perform quantitative hCG test 10 days or 13 days after S5 or S3 embryo transfer: (1) If there is a positive hCG test (>5 mIU/ml), the pregnancy will continue to be monitored; (2) Negative hCG test (<5 mIU/ml), we determined the outcome to be a failure in the first embryo transfer, and the study ended.

#### Cancel cycles

The cycle is canceled for COS cycles where no follicles are larger than 12 mm after ten days of ovarian stimulation. The characteristics of the canceled cycle (starting dose, total gonadotropin doses, COS days, LH, E2, and P4 measurements) are still recorded in the data collection table. The patient will have COS performed again in the next cycle.

#### Safety endpoints

The safety endpoints include the incidence of moderate or severe OHSS, miscarriage rates, ectopic pregnancy, and the complications of oocyte retrieval. Ovarian hyperstimulation syndrome (OHSS) is due to the excessive response of the ovaries to ovarian stimulation. OHSS is an uncommon complication (1 - 5% per cycle) and dangerous during ovarian stimulation. According to the American Society for Reproductive Medicine (ASRM) in 2016, OHSS is commonly classified into mild, moderate, severe, and critical based on symptoms, ovarian size, ascites, and haemoconcentration (Hct). Mild OHSS is diagnosed when presenting abdominal bloating, mild abdominal pain, and ovarian size < 8cm. Moderate OHSS is diagnosed by the ultrasonographic presence of ascites, ovarian size of 8-12 cm, with Hct >41%, and increased white blood cell count (>15 x  $10^9$ /L). Severe OHSS is defined as clinical ascites (occasionally pleural effusions), Oliguria, hematocrit>45%, hypoproteinemia, and ovarian size usually >12 cm. Critical OHSS is diagnosed by tense ascites or large pleural effusions, hematocrit>55%, white blood cell count >25 x 10<sup>9</sup>/L, oliguria/anuria, thromboembolism, acute respiratory distress syndrome, and so on. Complications of oocyte retrieval: (1) Vaginal bleeding: After completing the oocyte retrieval, the patient will have a speculum placed to examine the vagina. If bleeding is seen at the needle puncture site, the clinician will use gauze to press on the bleeding site and wait about 5 minutes. After that, the clinician checks again; if there is still bleeding, the clinician will sew the needle puncture site. (2) Bladder hemorrhage: caused by the needle piercing the egg through the bladder, with the primary symptom being red urine. Most cases will not require intervention. Patients should drink plenty of water, and in some cases, hemostatic drugs or antibiotics may be considered. If red urine persists or has blood clots in the bladder, washing the bladder could be regarded, and a cystoscopy could be performed to stop the bleeding. (3) Internal bleeding due to ovarian cyst rupture: After oocyte retrieval, if the patient has symptoms: abdominal pain (lower abdomen, one side or both sides, can spread to the shoulders), abdominal examination shows tenderness and reflexes abdominal wall, pain when touch pouch of Douglas or lethargy, fatigue, pale skin. The patient will be monitored for vital signs (pulse, blood pressure, temperature, SpO2),

and an ultrasound will be performed to check the ovaries, fluids, and abdominal cavity. At

the same time, we will take blood to test for red blood cell index, hemoglobin, and

hematocrit. If the patient's vital signs are stable, the amount of abdominal fluid is low, and

the hematocrit is > 30%, the patient will be using hemostatic medication; the vital signs

and hematocrit are monitored to determine whether the bleeding continues. When there are

hemodynamic changes, or the hematocrit continues to decrease below 30%, the patient

undergoes laparoscopic surgery to find the bleeding site in the ovary and cauterize the

bleeding. (4) Infection at the egg retrieval site: infrequent, with symptoms such as fever,

lower abdominal pain, pain on one side of the pelvis with increased white blood cells, and

increased CRP. The patient will be treated with broad-spectrum antibiotics according to

the hospital protocol.

The method of data collection

Personnel: This includes one main researcher and three associates.

*Tools:* Conducted using data collection table (Appendix 1)

Data collection plan: The data collection process corresponding to each step of the

research process, shown in detail in Figure 2.3, is expected to occur over 18 months

(from January 1, 2023, to June 30, 2024).

Research variables

Independent variable

**Table 1 Independent variables** 

| Variable name | Define | Туре | Scale/encoding | Unit | How to collect |
|---|---|---|---|---|---|
| Treatment grouping | One of 2 groups: Intervention group: using PPOS protocol. Control group: using GnRH-ant regimen | Qualitative,<br>binary | 0 = control group (GnRH-ant regimen) 1 = Intervention group (PPOS regimen). | | According to medical records |
| Time | Time point for LH quantification | Discrete qualitative | 1 = S6 $2 = S8$ $3 = ovulation day$ | | According to medical records |
| Sampling location | Center/hospital where samples were collected. There is significant clustering of the data and may contribute to random effects on the observed results. | Discrete<br>qualitative | 1,2,3: number corresponding to each hospital/reproduction center | | |

#### **Covariations**

#### **Table 2 Covariates**

| Variable<br>name | Define | Туре | Scale/encoding | Unit | How to collect |
|---|---|---|---|---|---|
| | A. Cha | racteristics of t | he study populatio | on | |
| Age | Time is calculated in calendar years from the date of birth on the wife's ID card to the date of participation in the study | Continuous variables | [20 – 45] | Years | Administrative information from medical records |
| Height | Height at the time of selection for the study, accurate to 0.5 cm | Continuous dosing | [150, 165.5,<br>172] | cm | Direct<br>measurement |
| Weight | Body weight<br>at the time of<br>selection for<br>the study | Continuous variables | [45, 55 60] | kg | Direct<br>measurement |

| Variable<br>name | Define | Туре | Scale/encoding | Unit | How to collect |
|---|---|---|---|---|---|
| BMI | The patient's body mass index, according to the formula: BMI=Weight (kg)Height (m)2 | Continuous variables | [19.1 23.4] | kg/m² | Secondary data, calculated from height and weight |
| Infertility period | Time from when you wanted to have a baby and did not use contraceptives until you were selected for the study | Continuous variables | [twelfth] | month | Interview and record in medical records |
| Causes of infertility | Is the cause of<br>the patient's<br>infertility | Identification | <ul><li>0 = Male factor</li><li>1 = Fallopian</li><li>tube factor</li></ul> | | Based on diagnosis recorded in |

| Variable<br>name | Define | Туре | Scale/encoding | Unit | How to collect |
|---|---|---|---|---|---|
| AFC | Number of | Discrete | 2 = POR 3 = Ovulatory disorders 4 = Unknown cause | ovarian | medical records Test |
| | ovarian follicles measuring 2 - 10mm on transvaginal ultrasound on day 2 of the menstrual cycle | quantification | | follicles | results/medical records |
| AMH | Patient's AMH concentration before IVF (up to 3 months) | Quantitative, continuous | [0.5,1,2,] | ng/ml | Test results/medical records |

| Variable<br>name | Define | Туре | Scale/encoding | Unit | How to collect |
|---|---|---|---|---|---|
| | B. Charact | teristics of the in | ı vitro fertilization | cycle | |
| Gonadotropin starting dose | The first dose of gonadotropin (FSH + hMG) is administered during the ovarian stimulation cycle | Identification | <ol> <li>0. 150</li> <li>1. 225</li> <li>2. 300</li> <li>3. 375</li> </ol> | IU | Take notes from medical records |
| Total<br>gonadotropin<br>dose | Total number of FSH + hMG drug units injected for ovarian stimulation | Quantitative, continuous | [1800,] | IU | Take notes from medical records |
| COS time | Number of<br>days of FSH +<br>hMG<br>injection | Quantitative, continuous | [8,] | day | Take notes<br>from medical<br>records |

| Variable<br>name | Define | Туре | Scale/encoding | Unit | How to collect |
|---|---|---|---|---|---|
| Number of<br>days using<br>GnRH-ant | Actual number of days of GnRH-ant use in the GnRH- ant subgroup. | Quantitative, continuous | [4,] | day | Take notes from medical records |

## Primary outcomes of the study (dependent variable)

## **Table 3 Dependent variables in the study**

| Variable name | Define | Туре | Scale/encoding | Unit | How to collect |
|---|---|---|---|---|---|
| | A. 0 | varian stimula | tion results | | |
| Expected number of oocytes | Expected number of oocytes to be collected: number of oocytes with size ≥ 12 mm on the day of ovulation. | Quantitative, discrete | [0,1,2,3] | oocytes | Recorded from medical records |
| Number of oocytes obtained | | Quantitative, discrete | [0,1,2,3] | oocytes | Recorded from |

| Variable name | Define | Туре | Scale/encoding | Unit | How to collect |
|---|---|---|---|---|---|
| | after aspiration under the guidance of transvaginal ultrasound. | | | | medical records |
| Number of MII oocytes | Number of ovarian follicles at metaphase II (MII) stage obtained after aspiration under the guidance of a transvaginal ultrasound probe | Quantitative, discrete | [0,1,2,3] | oocytes | Recorded from medical records |
| Number of fertilized oocytes | Number of oocytes with 2 pronuclei appearing after about 18-20 hours after performing ICSI | Quantitative, discrete | [0,1,2,3] | oocytes | Recorded from medical records |

| Variable name | Define | Туре | Scale/encoding | Unit | How to collect |
|---|---|---|---|---|---|
| Number of embryos N3 | Number of N3 embryos obtained after fertilization | Quantitative, discrete | [0,1,2,3] | Embryo | Recorded from medical records |
| Number of embryos N5 | Number of N5<br>embryos<br>obtained after<br>fertilization | Quantitative, discrete | [0,1,2,3] | Embryo | Recorded from medical records |
| No embryos | The condition of eggs not being able to create embryos after IVF/ICSI | Binary | 0 = No $1 = Yes$ | | Recorded from medical records |
| Cancel cycle | The COS cycle is canceled according to the criteria in section 2.5.3 | Binary | 0 = No<br>1 = Yes | | Recorded from medical records |
| Ovarian hyperstimulation (OHSS) | Is a treatment-induced complication of | Binary | 0 = No<br>1 = Yes | | Monitor and record from |

| Variable name | Define | Туре | Scale/encoding | Unit | How to collect |
|---|---|---|---|---|---|
| | physiological ovarian hyperstimulation, characterized by symptoms of varying degrees as described in section 2.6. | | | | medical records |
| OHSS level | The severity of OHSS is classified according to the standards in section 2.6 | Qualitative | 0 = Mild<br>1 = Average<br>2 = Severe<br>3 = Critical | | Monitor and record from medical records |
| | B. Describe | the progressio | n of LH hormone | | |
| Average LH concentration | LH concentration was measured repeatedly on days S6, S8 and the day to initiate oocyte | Quantitative, continuous | [ 1,1 ] | IU/L | Recorded from medical records |

| Variable name | Define | Туре | Scale/encoding | Unit | How to collect |
|---|---|---|---|---|---|
| | maturation and induce ovulation. | | | | |

Note: From these primary variables, secondary outcomes can be determined, for example: ratio of MII oocytes / total number of aspirated oocytes; ratio of retrieved oocytes/expected total number of oocytes; ratio of fertilized oocytes/total number of oocytes collected, etc.

#### Statistical analysis plan

Data analysis and visualization were done using the R programming language (ver 4.3.1). The following analytic procedure was applied to evaluate multiple outcomes across successive stages of a controlled ovarian stimulation procedure: (1) For the count data outcomes, such as the number of retrieved oocytes and number of maturated (MII) oocytes, their distribution was described using median and 5th to 95th percentiles. The adjusted effect of the PPOS regimen on these outcomes will be evaluated by a Negative Binomial (NBI) regression analysis; (2) The success rates, including maturation rate, fertilization rate, probabilities of achieving Day 3 and Day 5 embryos, as well as their transferability, were also described as median and 5th to 95th percentiles. The effectiveness of the PPOS protocol compared to GnRH-ant on the probability of success was evaluated as adjusted risk difference (aRD) and odds ratio (aOR) via a binomial regression model; (3) To achieve a precise estimation of the PPOS protocol's effect, adjustment for multiple baseline and procedural factors such as maternal age, AFC, baseline levels of AMH, LH, trigger method,

total FSH dose and length of stimulation was applied to regression analysis. The plausibility of each adjusted factor was confirmed based on data visualization and statistical analysis of the relationship between that factor and the targeted outcome. NBI and binomial regression models were fitted using the GAMLSS package (18). Confidence intervals for the marginal effects were determined by the delta method (19). Statistical inferences were based on null hypothesis testing at the significance level 0.05.

#### ETHICS IN RESEARCH

During IVF/ICSI, preventing premature luteinization is an essential part of COS ovarian stimulation. Among the current COS regimens, the antagonist COS regimen is the most commonly used regimen because it helps shorten ovarian stimulation time and is patientfriendly by reducing the amount of exogenous gonadotropin drugs required. injection and reduce treatment costs. However, the effectiveness in preventing LH surge is still quite variable. Recently, the PPOS regimen was born with the purpose of inhibiting the LH peak and preventing ovulation from occurring. Still, it has proven to be advantageous when the progestin route of administration is oral, meeting patient friendliness because of the reduction in the worry of having to inject too much medicine during the COS cycle. At the same time, progestin is also much cheaper than subcutaneous GnRH-ant. It should be noted that, until now, no regimen is optimal in effectiveness for all subjects. This also contributes to ensuring fairness and ethics in research. When participating in the study, patients are fully counseled about ovarian stimulation drugs, the IVF procedure, and the risks of complications that may occur during IVF, such as bleeding, vagina at the oocyte retrieval site, internal bleeding due to ovarian cyst rupture or infection at the aspiration site, ovarian hyperstimulation syndrome, possibility of cycle cancellation, fertilization rate, clinical pregnancy, and study progress (0. Patients also know which regimen they will use when undergoing ovarian stimulation (open-label). When agreeing to participate in the study, the patient will sign a consent form to participate in the study (04). All patient information is encrypted and confidential, used only for research purposes, not for any other purpose.

#### Patient and public involvement

Patients and the public are not involved in the trial process.

#### SUMMARY OF THE RESEARCH IMPLEMENTATION PROCESS

**Table 4 Summary of the research implementation process** 

| | Research stages | | | | | |
|---|---|---|---|---|---|---|
| Time | Sample selection | Random grouping | | After randomization | | |
| | After examination | Third day of menstruation | Ovarian<br>stimulation | Embryo<br>transfer | Monitor | |
| Sample selection | | | | | | |
| Receiving patients | X | | | | | |
| Examination | X | | | | | |
| Basic testing | X | | | | | |
| Sign consent | X | | | | | |
| Random grouping | | X | | | | |
| Intervention | | | | | | |
| PPOS regimen | | | x - | | | <b>→</b> |
| GnRH-anta regimen | | | X - | | | <b>→</b> |
| Sampling and outcome assessment | | | | | | |

| | Research stages | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Time | Sample selection | Random grouping | After randomization | | | | | After randomization |
| | After examination | Third day of menstruation | Ovarian<br>stimulation | Oocyte<br>aspiration | Fertilization<br>and embryo<br>culture | Embryo<br>transfer | Monitor | |
| Anthropometry and physiological status | x | | | | | | | |
| Characteristics of KTBT | | | x | | | | | |
| Main outcome | | | | | | | | |
| Pregnancy progresses | | | | | | | х | |
| Secondary<br>outcomes | | | | | | | | |
| Expected number of oocytes, number of oocytes recovered, number of MII oocytes, cycle cancellation Number of fertilized ovules, N3, N5 | | | | X | | | | |
| embryos, no<br>embryos | | | | | X | | | |
| OHSS | | | | X | | | | |

| | | | Research stages | | | | |
|---|---|---|---|---|---|---|---|
| Time | Sample<br>selection | Random<br>grouping | After randomization | | | | |
| | After examination | Third day of menstruation | Ovarian stimulation | Oocyte aspiration | Fertilization<br>and embryo<br>culture | Embryo<br>transfer | Monitor |
| Average LH concentration | | | х | | | | |

#### **FIGURE**



Figure 1 Results from the simulation estimate the sample size.

Note: According to this result, a sample comprising 200 patients (split equally between the groups) would be required. This size ensures that no difference in the number of retrieved or MII oocytes between the PPOS and control group would exceed 1.5 units.



Figure 2 Flowchart of the participant allocation

#### **APPENDIX**

#### **APPENDIX 1**

#### **DATA COLLECTION TABLE**

#### **STUDY**

# COMPARISON OF FERTILISATION RESULTS BETWEEN TWO OVARIAN STIMULATION PROTOCOLS WITH PROGESTIN AND ANTAGONIST IN VIETNAM POPULATION

# **DATA COLLECTION TABLE**

| I. PATIENT INFORMATION |
|-------------------------------------------------------------|
| Hospital: |
| File number: |
| First and last name: |
| Date of birth: [ ][ ] / [ ][ ] / [ ][ ][ ] (Day Month Year) |
| Phone number: |
| Phone number (husband or other relative): |
| PROTOCOL used: [ ] PPOS [ ] GnRH-ant |

#### II. DATA COLLECTION

#### A. BACKGROUND INFORMATION

| Code | Question | Reply | Note |
|------|---------------|-------|------|
| A1 | Date of birth | | |

| Code | Question | Reply | Note |
|---|---|---|---|
| | | Day month Year | |
| A2 | Height | [ ][ ][ ] cm | |
| A3 | Weight | [ ][ ],[ ]kg | |
| A4 | Infertility period | [ ][ ][ ] month | |
| A5 | Causes of infertility <sup>1</sup> | [] 0. Male factor [] 1. Fallopian tube factor [] 2. POR [] 3. PCOS [] 4. Unknown cause | |
| Day 2 - 3 of menstrual cycle | | | |
| A6 | AMH | [ ][ ],[ ] ng/ml | |
| <b>A7</b> | AFC <sup>2</sup> | [][] | |

#### **B. OVARIAN STIMULATION PROCESS**

(S1 start date: [ ][ ] / [ ][ ] / [ ][ ][ ][ ])

| Code | Question | Rep | | Note | |
|---|---|---|---|---|---|
| B1 | First dose of gonadotropins | [] 150 IU [] 225 IU [] 300 | | | |
| B2 | Day | E2 concentration (pg/ml) | P4 concentration (ng/ml) | LH | (IU/L) |

<sup>&</sup>lt;sup>1</sup>If multiple causes coexist, choose the most dominant cause

<sup>&</sup>lt;sup>2</sup>Ovarian follicle size 2 - 10 mm

| Code | Question | Repl | Reply |
|---|---|---|---|
| | [ ][ ] / [ ][ ]<br>(Day S6) | [ ][ ][ ][ ][ ]] | [ ][ ],[ ][ ] |
| | [ ][ ] / [ ][ ] (Day S8) | [ ][ ][ ][ ][ ] | [ ][ ],[ ][ ] |
| | [ ][ ] / [ ][ ]<br>(Trigger) | [ ][ ][ ][ ][ ] | [ ][ ],[ ][ ] |
| В3 | Total gonadotropin dose | [ ][ ][ ][ ] IU | |
| B4 | COS time | [ ][ ] day | |
| B5 | Number of days using GnRH-ant <sup>3</sup> | [ ][ ] day | |
| В6 | Early LH peak | [] 0. No [] 1. Yes (on date | |
| В7 | Number of cancellation cycles | [][] | |

#### **B'. OVARIAN STIMULATION PROCESS**

| (S1 start date: | [ | ][ | ] | / | [ ] | ][ | ] . | /[ | ][ | ][ | ][ | ]) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|---|---|---|

(For canceled cycles)

<sup>&</sup>lt;sup>3</sup>For the GnRH-ant protocol group

| Code | Question | | Reply | | | |
|---|---|---|---|---|---|---|
| B'1 | First dose of gonadotropins | | [] 150 IU [] 22. | | | |
| | Day | | pg/ml) P4 concentration (ng/ml) | | | ncentration |
| B'2 | [][]/[][]<br>(Day S6) | [][] | ][ ][ ],[ ][ ] | [ ][ ],[ ][ ] | [] | [],[][] |
| 52 | [][]/[][]<br>(Day S8) | [ ][ ][ ][ ][ ][ ] | | [ ][ ],[ ][ ] | [][],[][] | |
| | [ ][ ] / [ ][ ] (Trigger) | [ ][ ][ ][ ],[ ] | | [ ][ ],[ ][ ] | [] | [ ],[ ][ ] |
| В'3 | Total gonadotropin de | ose | [ ][ ][ ][ ] IU | | | |
| B'4 | COS time | | [ ][ ] day | | | |
| B'5 | Number of days using GnRH-<br>ant <sup>4</sup> | | [ ][ ] day | | | |
| B'6 | Early LH peak | | [] 0. No [] 1. Yes (on date) | | | |

#### C. RESULTS OF EMBRYORA AVOLUTION AND INFERTILATION

| (Date of oocyte retrieval [ ] | ][]/[][]/[][][] |
|-------------------------------|-----------------|
|-------------------------------|-----------------|

<sup>&</sup>lt;sup>4</sup>For the GnRH-ant regimen group

| Code | Question | Reply | Note |
|-----------|-----------------------------|-------|------|
| C1 | Expected number of oocytes | [][] | |
| C2 | Number of oocytes obtained | [][] | |
| С3 | Number of MII oocytes | [][] | |
| C4 | Number of fertilized ovules | [][] | |
| C5 | Number of blanks | [][] | |
| <b>C6</b> | Number of embryos N3 | [][] | |
| C7 | Number of embryos N5 | [][] | |

**APPENDIX 2** 

RESEARCH INFORMATION SHEET FOR PATIENTS

I. INFORMATION ABOUT RESEARCH

Study name: "COMPARISON OF FERTILISATION RESULTS BETWEEN TWO

**OVARIAN STIMULATION PROTOCOLS** WITH **PROGESTIN** AND

ANTAGONIST IN VIETNAM POPULATION."

Researcher and contact information

Main implementer: Doctor. Than Trong Thach

Contact phone: +84908.40.00.40

Email: thachthan007@gmail.com

Research sponsor: This research was not sponsored by any individual or entity. The

person conducting the research pays for the necessary expenses of the research

themselves.

II. RESEARCH PURPOSES

Progestin-primed ovarian stimulation regimen (using Dydrogesterone as a "primer" for

the COS cycle) compared to a conventional ovarian stimulation regimen (GnRH-ant and

gonadotropin) in Vietnamese women. performed in vitro fertilization.

III. REASON FOR INVITING TO PARTICIPATE IN THE STUDY

You were invited to participate in this study because you were treated with in vitro

fertilization and met the above study inclusion criteria. You need to carefully read and

understand the content provided in this information sheet. Before you decide to

participate in this study, you will be carefully explained about the research objectives and procedures, and you can also ask questions if necessary. After you are satisfied and understand this study and want to participate, you will sign a voluntary commitment to participate.

#### IV. RESEARCH PROCESS

#### **Step 1: Invite to participate in the study**

When you come for a check-up at the Artificial Reproductive Technology Center of Tam Anh General Hospital, Hanoi, the doctor will review the standards after performing basic surveys of the infertility examination process. receive and eliminate her. If you meet the sample selection criteria, your doctor will invite you to participate, advise you on the research process, the benefits and risks of participating, and answer your questions. If you agree to participate, you will sign consent to participate in the study.

#### **Step 2: Randomize groups**

After signing consent to participate in the study, she will be randomly assigned to 1 of 2 study subgroups (PPOS regimen group or GnRH-ant regimen group). You will know which group you are in. The doctor will collect some of your information into a data collection table.

#### Step 3: Stimulate the ovaries and monitor follicle development

First, you will be injected with ovarian stimulation medication starting on the 2nd or 3rd day of your menstrual cycle (called stimulation day S1). From day 5 onwards, the doctor will adjust or maintain the drug dose according to the response of the ovaries until ovulation is stimulated. The doctor will monitor the response of the ovaries by transvaginal ultrasound to measure the size of ovarian follicles, and the concentration of estradiol (E2), LH, and progesterone (P4) in the serum will be measured on the morning

of S5, S8, and ovulation induction day. To prevent a premature LH peak, for **the GnRH-anta protocol**, you will receive a subcutaneous injection of 0.25 mg of Cetrorelix (Cetrotide; Merck Serono) once daily from S5, along with ovarian stimulation medication until the day before. when ovulation is triggered. For **the PPOS protocol**, she will receive Dydrogesterone (DYG) 10mg, 1 pill x 3 times/day from S1 and continuously every day until the day of oocyte retrieval. When there are more than 2 ovarian follicles with a diameter greater than 17 mm, she will inject oocyte maturation medication with Triptoreline 0.2mg (Diphereline; Ipsen) or hCG 10,000 IU (IVF C 5000; LG) or recombinant hCG DNA 250 mcg (Ovitrelle; Merck Serono), and oocyte retrieval was performed 36 – 38 hours later. For stimulation cycles where no follicles are larger than 15 mm after 7 days of ovarian stimulation, the cycle is canceled. She will still have ovarian stimulation done again in the next cycle.

#### Step 4: Oocyte retrieval, fertilization, and embryo culture

The doctor will perform transvaginal oocyte retrieval 36 - 38 hours after the injection of medication to trigger oocyte maturation. After aspiration, the eggs will be fertilized by intracytoplasmic sperm injection (ICSI). Embryos will be cultured until day 3 or day 5 (depending on the number of embryos and the clinician's decision) and then completely frozen.

#### **Step 5: Monitor the patient after oocyte retrieval**

After aspiration, you will be monitored and treated for the following complications. These are complications that can occur with any IVF process.

- Vaginal bleeding: After the oocyte retrieval is completed, a speculum will be placed to examine the vagina. If bleeding is seen at the needle puncture site, the doctor will use gauze to press on the bleeding site and wait for a while. 5 minutes. After that,

the doctor checks again, and if there is still bleeding, he can consider injecting hemostatic medicine.

- Bladder hemorrhage rarely occurs due to the needle piercing the egg through the bladder, with the main symptom being red urine. Most cases will not require intervention. You will be told to drink plenty of water, and in some cases, hemostatic medication or antibiotics may be considered. If red urine persists or there are blood clots in the bladder, bladder irrigation, and cystoscopy can be performed to stop the bleeding.
- Internal bleeding due to ovarian cyst rupture: After oocyte retrieval, if there are symptoms of abdominal pain (lower abdomen, one side or both sides, can spread to the shoulders), lethargy, or fatigue, you will be examined and Perform tests to diagnose. Subsequent treatment will be performed according to the hospital's protocol.
- Infection at the egg retrieval site: very rare, with symptoms such as fever, lower abdominal pain, and pain on one side of the pelvis, and blood tests are performed to determine infection. After that, she will be treated with broad-spectrum antibiotics according to the hospital protocol.
- Ovarian hyperstimulation syndrome is due to excessive response of the ovaries to ovarian stimulation. This is an uncommon complication (1 5% in one cycle) but is a dangerous complication during ovarian stimulation. You may have symptoms such as abdominal pain, nausea, vomiting, difficulty breathing, rapid weight gain, and decreased urination. Depending on the level of symptoms and tests, it can be divided into levels: mild, moderate, severe and critical; and she will be monitored and treated according to the hospital's protocol.

#### **Step 6: Embryo transfer and confirmation of pregnancy**

You will have frozen embryos transferred in the next cycle and a quantitative hCG test will be performed 10 days or 13 days after N5 or N3 embryo transfer: (1) If the hCG test is positive (> 5 mIU/ml), the pregnancy will continue to be monitored; (2) If the hCG

test is negative (< 5mIU/ml), the outcome is determined as failure in the first embryo transfer and the study ends. She will still continue to undergo IVF according to the hospital's protocol.

# V. RESPONSIBILITIES OF RESEARCH SUBJECTS WHEN PARTICIPATING IN RESEARCH

You need to follow the instructions of your doctor and midwife and complete all steps in the treatment and research process as described above because of the study's possible risks and side effects. When performing IVF, you will have risks and side effects of IVF treatment, such as:

- 1) Complications of the oocyte retrieval process, such as vaginal bleeding, internal bleeding due to ovarian cyst rupture, bladder bleeding, and infection at the retrieval site: rarely occur; you will be evaluated by a doctor. , monitor and treat if there is a risk or this condition occurs as in step 5 of the research process
- 2) Ovarian hyperstimulation is when the ovaries respond greatly to ovarian stimulation drugs. Ovarian hyperstimulation can cause bloating, abdominal pain, and polymembranous effusion. Your doctor will evaluate your condition, monitor and treat you if there is a risk or this condition occurs, as in step 5 of the research process.
- 3) Cycle cancellation: a condition in which no ovarian follicles are larger than 12 mm after ten days of ovarian stimulation. Your condition will be evaluated with canceled cycles, and your ovaries will be stimulated again in the next cycle.
- 4) Embryo transfer but negative pregnancy test results: due to the nature of the study, only data is recorded on the first embryo transfer, so if the pregnancy test result is negative, the study will end, but you will still be able to continue fertilization treatment. Test tube sperm according to hospital protocol.

#### VII. BENEFITS OF PARTICIPATING IN RESEARCH

You will be thoroughly explained and monitored throughout the in vitro fertilization treatment process.

#### VIII. INFORMATION SECURITY

Your information will be kept confidential in your medical record. When collecting data, all personal information will be encrypted, stored separately, and used only for research purposes.

#### IX. DO NOT PARTICIPATE IN RESEARCH

The choice to participate in the study is yours and voluntary. If you have been accepted into the study but change your mind, you can withdraw from the study at any time. She will still be cared for and treated like a routine in vitro fertilization case.

#### X. COSTS OF TREATMENT AND COSTS OF RESEARCH

You will not be paid for participating in the research. You will still pay the cost of COS injections and the cost of performing in vitro fertilization as in normal treatment cases, according to hospital regulations.

#### XI. CONTACT

If you have any questions about the study, please contact Dr. Than Trong Thach at +84908 400 040 or by email at thachthan007@gmail.com.

**APPENDIX 3** 

CONSENT TO PARTICIPATE IN RESEARCH

Research name

"COMPARISON OF FERTILISATION RESULTS BETWEEN TWO OVARIAN

STIMULATION PROTOCOLS WITH PROGESTIN AND ANTAGONIST IN

VIETNAM POPULATION. "

Researcher and contact information

Main researcher: Dr. Than Trong Thach

Contact Phone: +84908.40.00.40

Email: thachthan007@gmail.com

I voluntarily participated in this study. I have read and clearly understood the purpose and

procedure of the research. The study was explained clearly; I had time to ask questions

about the study, and I was satisfied with all the answers.

Name of study participant

Signature

Date

Confirmation of the person conducting the research

| I, the undersigned, commit to fully explaini<br>and ensuring that research participants cle | | 1 1 |
|---|---|---|
| and benefits of participating in the study. | _ | |
| Name of person conducting research | Signature | Date |

#### **REFERENCES**

- 1. Bosch E, Valencia I, Escudero E, Crespo J, Simón C, Remohí J, Pellicer A. Premature luteinization during gonadotropin-releasing hormone antagonist cycles and its relationship with in vitro fertilization outcome. Elsevier Inc.; 2003. p. 1444-9.
- 2. Macklon NS, Stouffer RL, Giudice LC, Fauser BCJM. The Science behind 25 Years of Ovarian Stimulation for in Vitro Fertilization. Oxford Academic; 2006. p. 170-207.
- 3. Kuang Y, Chen Q, Fu Y, Wang Y, Hong Q, Lyu Q, et al. Medroxyprogesterone acetate is an effective oral alternative for preventing premature luteinizing hormone surges in women undergoing controlled ovarian hyperstimulation for in vitro fertilization. Fertil Steril; 2015. p. 62-70.e3.
- 4. Yu S, Long H, Ya-Ning Chang H, Liu Y, Gao H, Zhu J, et al. New application of dydrogesterone as a part of a progestin-primed ovarian stimulation protocol for IVF: a randomized controlled trial including 516 first IVF/ICSI cycles. Hum Reprod; 2018. p. 229-37.
- 5. Xiao Zn, Peng Jl, Yang J, Xu Wm. Flexible GnRH Antagonist Protocol versus Progestin-primed Ovarian Stimulation (PPOS) Protocol in Patients with Polycystic Ovary Syndrome: Comparison of Clinical Outcomes and Ovarian Response. Huazhong University of Science and Technology; 2019. p. 431-6.
- 6. Wang N, Zhu Q, Ma M, Liang Z, Tao Y, Wang Y, Kuang Y. Comparison of a progestin-primed ovarian stimulation protocol with a flexible GnRH antagonist protocol in patients with polycystic ovary syndrome who are participating in an IVF programme: study protocol for a randomised controlled trial. BMJ Open. 2020;10(12):e038153.
- 7. Chen Q, Chai W, Wang Y, Cai R, Zhang S, Lu X, et al. Progestin vs. Gonadotropin-Releasing Hormone Antagonist for the Prevention of Premature Luteinizing Hormone Surges in Poor Responders Undergoing in vitro Fertilization Treatment: A Randomized Controlled Trial. Front Endocrinol (Lausanne); 2019.

- 8. Du M, Zhang J, Li Z, Liu X, Li J, Liu W, Guan Y. Comparison of the Cumulative Live Birth Rates of Progestin-Primed Ovarian Stimulation and Flexible GnRH Antagonist Protocols in Patients With Low Prognosis. Frontiers Media S.A.; 2021. p. 1155.
- 9. Guo Yc, Chen Py, Li Tt, Jia L, Sun P, Zhu Ws, et al. Different progestin-primed ovarian stimulation protocols in infertile women undergoing in vitro fertilization/intracytoplasmic sperm injection: an analysis of 1188 cycles. Springer Verlag; 2019. p. 1201-12.
- 10. Gurbuz AS, Gode F. Dydrogesterone-primed ovarian stimulation is an effective alternative to gonadotropin-releasing hormone antagonist protocol for freeze-all cycles in polycystic ovary syndrome. Journal of Obstetrics and Gynaecology Research. 2020;46(8):1403-11.
- 11. Chen Q, Wang Y, Sun L, Zhang S, Chai W, Hong Q, et al. Controlled ovulation of the dominant follicle using progestin in minimal stimulation in poor responders. Reprod Biol Endocrinol; 2017.
- 12. Dozortsev D, Pellicer A, Diamond MP. Progesterone is a physiological trigger of ovulatory gonadotropins. Fertil Steril; 2020. p. 923-4.
- 13. Heikinheimo O, Gordon K, Williams RF, Hodgen GD. Inhibition of ovulation by progestin analogs (agonists vs antagonists): Preliminary evidence for different sites and mechanisms of actions. Elsevier; 1996. p. 55-64.
- 14. Griesinger G, Tournaye H, Macklon N, Petraglia F, Arck P, Blockeel C, et al. Dydrogesterone: pharmacological profile and mechanism of action as luteal phase support in assisted reproduction. Reproductive BioMedicine Online. 2019;38(2):249-59.
- 15. Rižner TL, Brožič P, Doucette C, Turek-Etienne T, Müller-Vieira U, Sonneveld E, et al. Selectivity and potency of the retroprogesterone dydrogesterone in vitro. Steroids. 2011;76(6):607-15.
- 16. Stanczyk FZ, Hapgood JP, Winer S, Mishell Jr DR. Progestogens used in postmenopausal hormone therapy: differences in their pharmacological properties, intracellular actions, and clinical effects. Endocrine reviews. 2013;34(2):171-208.

- 17. Cundill B, Alexander ND. Sample size calculations for skewed distributions. BMC medical research methodology. 2015;15:1-9.
- 18. Stasinopoulos MD, Rigby RA, Heller GZ, Voudouris V, De Bastiani F. Flexible regression and smoothing: using GAMLSS in R: CRC Press; 2017.
- 19. Arel-Bundock V. Marginal effects: predictions, comparisons, slopes, marginal means, and hypothesis tests. R package version 0.9. 0. 2023.